CLINICAL TRIAL: NCT07317778
Title: Chemotherapy Combine With or Without Adebrelimab and Trastuzumab Rezetecan(SHR-A1811) as Neoadjuvant Therapy for Hormone Receptor Positive/HER2 Low Early Stage Breast Cancer: A Randomized Phase II Trial
Brief Title: Chemotherapy With or Without Adebrelimab and T-DXh as Neoadjuvant Therapy for HR+/HER2 Low Early Stage Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, YING FAN, professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-094
Record Dates: First submitted 2025-12-11; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); HR Positive/HER2 Low Breast Cancer
Keywords: SHR-A1811; adebrelimab; Trastuzumab Rezetecan; HR+/HER2-low; early stage breast cancer
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: SHR-A1811-EC + Adebrelimab (Experimental): 4 cycles of SHR-A1811 follow by 4 cycles of EC chemotherapy, with concurrent adebrelimab throughout all 8 cycles.
  Interventions: Drug: SHR-A1811; Drug: Adebrelimab (PD-L1 inhibitor); Drug: Anthracycline & Cyclophosphamide treatment scheme
- Arm 2: T-EC + Adebrelimab (Experimental): 4 cycles of taxane follow by 4 cycles of EC chemotherapy, with concurrent adebrelimab throughout all 8 cycles.
  Interventions: Drug: Adebrelimab (PD-L1 inhibitor); Drug: Taxane Chemotherapy; Drug: Anthracycline & Cyclophosphamide treatment scheme
- Arm 3: T-EC (Active Comparator): 4 cycles of taxane follow by 4 cycles of EC chemotherapy
  Interventions: Drug: Taxane Chemotherapy; Drug: Anthracycline & Cyclophosphamide treatment scheme

INTERVENTIONS:
Drug: SHR-A1811 — An anti-HER2 ADC injection, administered on day 1 of each cycle, with one cycle every 3 weeks. 4.8mg/kg or 5.6mg/kg IV, according to the outcomes of the safety run in process.
  Other Names: Trastuzumab Rezetecan; T-DXh
  Arms: Arm 1: SHR-A1811-EC + Adebrelimab
Drug: Adebrelimab (PD-L1 inhibitor) — A PD-L1 inhibitor, 1200mg IV, is administered on the 1st day of every 3 weeks cycle.
  Other Names: SHR-A1316
  Arms: Arm 1: SHR-A1811-EC + Adebrelimab; Arm 2: T-EC + Adebrelimab
Drug: Taxane Chemotherapy — Could be paclitaxel, docetaxel or Nab-paclitaxel, according to physician's choice.
  Arms: Arm 2: T-EC + Adebrelimab; Arm 3: T-EC
Drug: Anthracycline & Cyclophosphamide treatment scheme — Anthracycline usually use epirubicin, 90-100mg/m2, combine with Cyclophosphamide 600mg/m2, both use at day 1, every 3 weeks cycle.

SUMMARY:
The goal of this clinical trial is to learn if add SHR-A1811 and/or Adebrelimab on standard chemotherapy could further improve the pCR rate in HR+/HER2 low early stage breast cancer patients. It will also learn about the safety of these combination regimen. The main questions it aims to answer are:

Is Adebrelimab plus chemotherapy better than T-EC chemotherapy alone in neoadjuvant setting of HR+/HER2-low early stage population? Is SHR-A1811-EC plus Adebrelimab better than T-EC chemotherapy and/or Adebrelimab plus chemotherapy

Participants will:

Take 8 cycles of standard chemotherapy at day1, every 3 weeks cycle(standard care), or take 8 cycles of adebrelimab plus standard chemotherapy at day 1, every 3 weeks cycle(experimental 2), or take 4 cycles of SHR-A1811 and Adebrelimab at day 1, every 3 weeks cycle, then 4 cycles of adebrelimab plus EC chemotherapy at day 1, every 3 weeks cycke(experimental 1).

Visit the clinic once every 6 weeks at neoadjuvant period for tumor assessment. Take surgery after completion of 8 cycles of neoadjuvant therapy and assess the pathological response. Then, visit the clinic once every 12 weeks at first year and then every 6 months for tumor assessment.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score: 0-1;
* Pathologically confirmed invasive breast cancer, with tumor stage T1c-T2, cN1-2 or T3-4 cN0-2;
* HR positive/HER2 low expression(defined as HER2 IHC 1+/2+, FISH negative);
* Known PD-L1 expression status, or sufficient tumor tissue for PD-L1 testing;
* Sufficient organ function
* Female patients who have not undergone menopause or sterilization, accept for abstain from sexual activity or use an effective contraceptive method during the treatment period and at least 7 months after the last administration of the study medication;
* Voluntarily participate and sign the informed consent form.

Exclusion Criteria:

* Inflammatory breast cancer;
* Previously received anti-tumor therapy or radiotherapy for any malignant tumor(not including cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma);
* Concurrently received anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy;
* Within 4 weeks before enrollment, underwent major surgical procedures unrelated to breast cancer, or the patient has not fully recovered from such procedures;
* Had clinically significant pulmonary diseases, including but not limited to interstitial pneumonia, pneumonia, pulmonary fibrosis and radiation pneumonia (except for radiological changes that do not require treatment), or was found to have such diseases during the screening period;
* Had any cardiac diseases, including: (1) Severe / unstable angina pectoris; (2) Requires drug treatment or has clinically significant arrhythmia; (3) Had a myocardial infarction within 6 months before enrollment; (4) Has symptomatic congestive heart failure with NYHA grade ≥ II; (5) Any other heart diseases judged by the researcher as not suitable for participation in this trial;
* Known to have had an allergic history to the components of the drug in this protocol; have a history of immunodeficiency, including positive HIV test, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation;
* Had severe comorbidities or other conditions that would interfere with the planned treatment, or any other situation that the researcher considered the patient was not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-10-15 (Estimated); Study Completion 2033-09-15 (Estimated)

PRIMARY OUTCOMES:
tpCR(ypT0/Tis ypN0M0) | After surgery (within 1 month)
  total pathological complete response, define as ypT0/Tis ypN0 M0 assessed according to the AJCC staging criteria

SECONDARY OUTCOMES:
EFS | from enrollment to completion of 3 years of follow up after surgery
  event free survival, defined as the time from randomization to disease progression that precluded surgery, local or distant recurrence, second primary cancer or death due to any cause, whichever occurred first.
OS | from enrollment to complete of 5 years follow up after surgery
  overall survival, define as the time from randomization to death due to any cause.
Adverse Events | AEs were assessed from enrollment throughout the trial and for 30 days after discontinuation of treatment (90 days for serious AEs)
  The safety assessment includes the categories and incidence rates of adverse events, as well as the severity grade according to CTCAE 6.0

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China